CLINICAL TRIAL: NCT02731326
Title: iPhone Helping Evaluate Atrial Fibrillation Rhythm Through Technology
Acronym: iHEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Suzanne Bakken, Alumni Professor of the School of Nursing, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAAO2555
Record Dates: First submitted 2016-03-24; First posted 2016-04-07 (Estimated); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- iHEART (Experimental): Participants will transmit daily ECGs using AliveCor for 6 months following cardioversion or ablation procedure to treat AF/AFL. Participants will also receive read-only behavioral altering messaging three times per week focusing on AF, cardiovascular risk factors, and healthy living.
  Interventions: Device: AliveCor; Behavioral: Behavioral Altering Messaging
- Usual Care (No Intervention): Participants will continue with usual care with their physician.

INTERVENTIONS:
Device: AliveCor — The AliveCor Heart Monitor, an FDA-approved smartphone technology, snaps on to the patient's study smartphone similar to a protective case and works through a free application, "AliveECG". It captures a highly sensitive (98%), specific (97%), and accurate (97%) single-lead ECG recording through two electrodes on the back of the patient's smartphone. When the application is opened, recording begins automatically when both electrodes make contact with skin. Transmissions are automatically uploaded to the study patient portal within the AliveCor "cloud".
  Arms: iHEART
Behavioral: Behavioral Altering Messaging — Behavioral altering messages relating to the participant's AF and underlying cardiac risk factors will be systematically selected from a bank of text messages developed through collaboration by the study team and an expert interdisciplinary panel from the American Heart Association. The content of the text messages will not include PHI. The final text message bank will be housed internally and maintained by the Data Manager and text messages will be pushed automatically from this database. The only identifying link to participants included in this database will be their study-provided phone number
  Arms: iHEART

SUMMARY:
Atrial fibrillation (AF), a condition where the top chambers of the heart beat irregularly, is a major health problem. The long-term goal of this project is to use a personal, mobile heart monitor to help patients better recognize recurrent AF and improve patients' ability to better manage their condition. A total of 300 patients with a history of AF will be included in the study, with 150 patients receiving an iPhone with the mobile monitoring device and educational text messaging and the remaining 150 patients continuing with their regular medical care. Each patient will be included in the intervention period for 6 months. The rate of recurrent AF and treatments meant to manage AF and other heart conditions will be determined for both groups. Patients in both groups will complete a series of questionnaires at the start and end of the 6 month study period to look at differences in quality of life and knowledge of AF.

DETAILED DESCRIPTION:
This study is a prospective randomized control trial with 1:1 randomization of 300 patients to either use the AliveCor device and receive behavioral altering motivational text messaging OR continue with usual care. The sample size and power was based on the test of the difference in AF detection rates between the intervention group and the control group in a similarly design pilot study. In the preliminary data there were 4 episodes of AF during the follow-up of 12 patients or a detection rate of 0.33 vs. a detection rate of 8% among controls. The detection window in this study as the time period from randomization to the 6-month follow-up will be defined. All patients' clinical records will be reviewed every month (via charts and/or internal and external electronic medical record systems) up until month 6 for initiations/changes in treatments targeting AF. A recurrence of AF in the chart and any related therapies that are initiated as a result of electrocardiogram (ECG) findings through usual cardiac care or from the AliveCor™ Heart Monitor will be specifically looked at. Changes in cardiovascular measures (blood pressure, glucose control, etc.) will be compared between groups. The effect of participating in the intervention, which includes targeted text messaging on AF knowledge and cardiovascular behavior change will be determined by comparing the change in AF knowledge scales from baseline to 6 months. This study will also measure and compare the incidence of documented AF in both groups, changes in prescribed treatment by healthcare providers over the 6-month period, and the relationship of the intervention to changes in cardiac measures and quality-adjusted life-years (QALYs) measured at baseline and 6 months. A biannual time period was chosen to capture AF redetection, changes in AF treatment, and self-reported quality of life based on other studies that have shown biannual time-points as most appropriate for collecting the proposed study endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Males and females (English or Spanish speaking) age ≥ 18 years with a history of AF in the last 30 days that was treated with normal rhythm restored.
* Ability to successfully use the AliveCor™ Heart Monitor, capture a baseline ECG, and transmit on the day of enrollment
* Demonstrated ability to receive, read, and send a text messages on the day of enrollment
* Willingness to complete the study questionnaires at baseline and 6 months

Exclusion Criteria:

* Documented permanent (chronic) AF
* Patient found to be in AF or other rhythm disturbances on the day of enrollment (i.e., they need to be clinically evaluated or treated)
* Unwillingness have their clinical data collected over the study period
* Unwillingness to receive and read cardiovascular text messaging three times a week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Bakken, PhD, RN, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Research data will be disseminated for the whole study sample and not individually.

REFERENCES:
- [Background] Hickey KT. Developing and Sustaining a Career as a Transdisciplinary Nurse Scientist. J Nurs Scholarsh. 2018 Jan;50(1):20-27. doi: 10.1111/jnu.12359. Epub 2017 Nov 14. PMID 29135066
- [Background] Hickey KT, Hauser NR, Valente LE, Riga TC, Frulla AP, Masterson Creber R, Whang W, Garan H, Jia H, Sciacca RR, Wang DY. A single-center randomized, controlled trial investigating the efficacy of a mHealth ECG technology intervention to improve the detection of atrial fibrillation: the iHEART study protocol. BMC Cardiovasc Disord. 2016 Jul 16;16:152. doi: 10.1186/s12872-016-0327-y. PMID 27422639
- [Background] Hickey KT, Riga TC, Mitha SA, Reading MJ. Detection and management of atrial fibrillation using remote monitoring. Nurse Pract. 2018 Mar 12;43(3):24-30. doi: 10.1097/01.NPR.0000530214.17031.45. PMID 29438185
- [Background] Hickey KT, Wan E, Garan H, Biviano AB, Morrow JP, Sciacca RR, Reading M, Koleck TA, Caceres B, Zhang Y, Goldenthal I, Riga TC, Masterson Creber R. A Nurse-led Approach to Improving Cardiac Lifestyle Modification in an Atrial Fibrillation Population. J Innov Card Rhythm Manag. 2019 Sep 15;10(9):3826-3835. doi: 10.19102/icrm.2019.100902. eCollection 2019 Sep. PMID 32494426
- [Result] Reading M, Baik D, Beauchemin M, Hickey KT, Merrill JA. Factors Influencing Sustained Engagement with ECG Self-Monitoring: Perspectives from Patients and Health Care Providers. Appl Clin Inform. 2018 Oct;9(4):772-781. doi: 10.1055/s-0038-1672138. Epub 2018 Oct 10. PMID 30304745
- [Result] Goldenthal IL, Sciacca RR, Riga T, Bakken S, Baumeister M, Biviano AB, Dizon JM, Wang D, Wang KC, Whang W, Hickey KT, Garan H. Recurrent atrial fibrillation/flutter detection after ablation or cardioversion using the AliveCor KardiaMobile device: iHEART results. J Cardiovasc Electrophysiol. 2019 Nov;30(11):2220-2228. doi: 10.1111/jce.14160. Epub 2019 Sep 25. PMID 31507001
- [Result] Koleck TA, Mitha SA, Biviano A, Caceres BA, Corwin EJ, Goldenthal I, Creber RM, Turchioe MR, Hickey KT, Bakken S. Exploring Depressive Symptoms and Anxiety Among Patients With Atrial Fibrillation and/or Flutter at the Time of Cardioversion or Ablation. J Cardiovasc Nurs. 2021 Sep-Oct 01;36(5):470-481. doi: 10.1097/JCN.0000000000000723. PMID 32675627
- [Result] Caceres BA, Hickey KT, Bakken SB, Biviano AB, Garan H, Goldenthal IL, Koleck TA, Masterson-Creber R, Turchioe MR, Jia H. Mobile Electrocardiogram Monitoring and Health-Related Quality of Life in Patients With Atrial Fibrillation: Findings From the iPhone Helping Evaluate Atrial Fibrillation Rhythm Through Technology (iHEART) Study. J Cardiovasc Nurs. 2020 Jul/Aug;35(4):327-336. doi: 10.1097/JCN.0000000000000646. PMID 32015256

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two individuals that were enrolled failed to convert to normal sinus rhythm during direct current cardioversion (DCCV) so became ineligible for the study after enrollment and consent. Only 262 out of 264 participants had their data collected and analyzed.
Groups:
- iHEART: Participants will transmit daily ECGs using AliveCor for 6 months following cardioversion or ablation procedure to treat AF/AFL. Participants will also receive read-only behavioral altering messaging three times per week focusing on AF, cardiovascular risk factors, and healthy living.
  AliveCor: The AliveCor Heart Monitor, an FDA-approved smartphone technology, works through a free application, "AliveECG". It captures a highly sensitive (98%), specific (97%), and accurate (97%) single-lead ECG recording through two electrodes on the back of the patient's smartphone. When the application is opened, recording begins automatically when both electrodes make contact with skin. Transmissions are automatically uploaded to the study patient portal within the AliveCor "cloud".
  Behavioral Altering Messaging: Behavioral altering messages relating to the participant's AF and underlying cardiac risk factors will be sent three times per week.
Period: Overall Study
Arm/Group | iHEART | Usual Care
Started | 131 | 131
Completed | 115 | 123
Not Completed | 16 | 8
Not completed — Withdrawal by Subject | 4 | 1
Not completed — No Cardioversion or Ablation Procedure | 1 | 6
Not completed — Discharged without AliveCor | 10 | 0
Not completed — Duplicate Participant | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | iHEART | Usual Care | Total
Number analyzed (Participants) | 115 | 123 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (12) | 61 (12) | 61 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 96 | 184
  Male | 27 | 27 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 17 | 27
  Not Hispanic or Latino | 61 | 67 | 128
  Unknown or Not Reported | 44 | 39 | 83
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 8 | 11
  White | 88 | 93 | 181
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 23 | 17 | 40
Region of Enrollment [Number; unit: participants]
  United States | 115 | 123 | 238
Procedure at Enrollment: Radiofrequency Ablation [Count of Participants; unit: Participants] | 60 | 43 | 103

OUTCOME MEASURES:

1. Primary Outcome: Rate of Recurrence of Atrial Arrhythmias
Description: Examine the rate of recurrent atrial arrhythmias between the intervention and control group during the study period. The investigators will define and calculate recurrent AF detection rate as the ratio of the number of recurrent AF episodes to the number of person-months of follow-ups.
Time Frame: Six months
Population: The analytic population excludes 5 individuals from the control group for whom we were unable to obtain follow-up data for this outcome variable. Data was collected and analyzed for 118 out of 123 participants in the Usual Care arm.
Measure: Mean (Standard Deviation); unit: episodes per person-month of follow-up
Arm/Group | iHEART | Usual Care
Number analyzed (Participants) | 115 | 118
episodes per person-month of follow-up | 0.132 (0.014) | 0.091 (0.012)
Statistical Analysis 1: Comparison: iHEART vs Usual Care; The study was designed to have 80% power to detect a hazard ratio of 2 for recurrence detection (α = .05). Kaplan-Meier curves were created for recurrence detection in the intervention and control groups over the 6-month follow-up period. Differences in time to recurrence between groups were assessed using a Cox proportional hazards model. Baseline variables that differed significantly between groups were included as covariates and adjusted Kaplan-Meier curves were constructed; Test type: Equivalence — The study was designed to have 80% power to detect a hazard ratio of 2 for recurrence detection (α = .05); p = 0.05, Regression, Cox; Hazard Ratio (HR) = 1.56, 95% CI 2-sided [1.06 to 2.30] — Treatment arm equals numerator. Control arm=denominator

2. Primary Outcome: Time to Treatment for Recurrence of Atrial Arrhythmia
Description: Time to treatment for recurrence of atrial arrhythmia from detection of arrhythmia to 6 months
Time Frame: Six months
Population: The analytic population only includes 58 out of 115 participants from the iHeart group and 49 out of 123 from the control group for whom we were unable to obtain data for this outcome variable.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | iHEART | Usual Care
Number analyzed (Participants) | 58 | 49
days | 43 (41) | 33 (36)
Statistical Analysis 1: Comparison: iHEART vs Usual Care; Kaplan-Meier curves were created for assessing time to treatment for intervention and control groups. Time to treatment was defined as the time interval from detection of a recurrent arrhythmia to treatment for that arrhythmia; Test type: Equivalence — The study was designed to have 80% power to detect a hazard ratio of 2 (α = .05); p = 0.05, Regression, Cox; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.09 to 0.58] — Treatment arm equals numerator. Control arm=denominator

3. Primary Outcome: Number of Intervention and Control Group Patients Treated for Recurrent Atrial Arrhythmia
Description: Number of intervention and control group patients with recurrent atrial arrhythmia who received treatment for recurrent atrial arrhythmia
Time Frame: 6 months
Population: The analysis population was the number of individuals who had recurrent atrial tachycardia detected in the intervention and control group. The analytic population only includes 58 out of 115 participants from the iHeart group and 49 out of 123 from the control group for whom we were unable to obtain follow-up data for this outcome variable.
Measure: Count of Participants; unit: Participants
Arm/Group | iHEART | Usual Care
Number analyzed (Participants) | 58 | 49
Participants | 21 | 35
Statistical Analysis 1: Comparison: iHEART vs Usual Care; Test type: Superiority; p < .0001, Regression, Cox; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.19 to 0.58]

4. Secondary Outcome: Difference in Quality-Adjusted Life Years (QALYS) Between Intervention and Control Groups
Description: The EQ-5D index is a summary measure that assesses the value for preferring one health state to another. The full range of the EQ-5D index is 0 to 1. The EQ-5D index is anchored at 0 for death and 1 for full (optimal) health, so that having a reduced score of 0.5 is equivalent to living in full health only 50% of the time. Therefore, one year lived at a reduced EQ-5D index of 0.5 equals 0.5 QALYs which is the same as living a half year in full health. Higher scores mean a better outcome. QALYs were calculated from baseline to six months for patients whose EQ-5D index scores were available at both baseline and follow-up.
Time Frame: Six Months
Population: The analysis population is the number of participants in the intervention and control group who had data on the EQ-5D at both baseline and follow-up which was required to calculate the QALYS. The analytic population only includes 58 out of 115 participants from the iHeart group and 56 out of 123 from the control group for whom we were unable to obtain follow-up data for this outcome variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iHEART | Usual Care
Number analyzed (Participants) | 58 | 56
score on a scale | 0.94 (0.14) | 0.91 (0.13)
Statistical Analysis 1: Comparison: iHEART vs Usual Care; Test type: Superiority; p = 0.24, t-test, 2 sided

5. Secondary Outcome: Change in Atrial Fibrillation Knowledge Scale (AFKS) Scores Between Baseline and Six Months
Description: Correlation between educational text messaging and participation in intervention on AF knowledge will be determined by comparing the change in mean scores between groups from the Atrial Fibrillation Knowledge Scale (AFKS) from baseline to 6 months. The AFKS is a valid instrument used to distinguish knowledge levels in AF patients. It is an 11-item scale including questions about AF in general, symptom recognition, and treatment and is validated (Cronbach α 0.58) to differentiate between knowledge changes in patients with AF. For each item patients can choose an answer out of three options, with one being the correct answer. The correct answer yields one point, while no points are added or subtracted to the score in case of an incorrect answer. The minimum score of the scale is 0 with a maximum score of 11.
Time Frame: Six months
Population: The analysis population comprised the participants who had complete data on the AFKS score at baseline and 6 months. The analytic population only includes 44 out of 115 participants from the iHeart group and 23 out of 123 from the control group for whom we were unable to obtain follow-up data for this outcome variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iHEART | Usual Care
Number analyzed (Participants) | 44 | 23
score on a scale | 0.27 (2.08) | .17 (2.93)
Statistical Analysis 1: Comparison: iHEART vs Usual Care; Test type: Superiority; p = 0.89, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months post enrollment procedure
Arm/Group | iHEART | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/131 | 0/131
Serious Adverse Events (participants affected / at risk) | 0/131 | 0/131
Other Adverse Events (participants affected / at risk) | 0/131 | 0/131

LIMITATIONS AND CAVEATS:
While there was primary outcome data for all participants with the exception of 5 in the control group, secondary outcome measures reflect less than half the participants in the intervention and control groups due to missing data. Thus, findings related to secondary outcome measures should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT02731326/Prot_SAP_000.pdf